CLINICAL TRIAL: NCT05161871
Title: Effectiveness of tDCS and Monoclonals Antibodies Anti-CGRP as a Combined Treatment for Migraine: a Randomized, Double-blind, Sham-controlled Trial
Brief Title: Transcranial Direct Current Stimulation Plus Monoclonal Antibodies Acting on the CGRP Pathway for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Simona Sacco, Full Professor of Neurology, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201722 ID INT 193/21
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cathodal transcranial direct current stimulation (Active Comparator)
  Interventions: Device: Cathodal transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator)
  Interventions: Device: Sham cathodal transcranial direct current stimulation

INTERVENTIONS:
Device: Cathodal transcranial direct current stimulation — The cathodal transcranial direct current stimulation protocol will consist in five daily sessions, each lasting 20 min. The montage will provide a bilateral stimulation on occipital areas, with the reference anodal electrodes positioned on the M1 areas. The stimulation will be applied via 4 conductive-rubber square electrodes (5x5 cm) placed in sponges saturated with high conductivity gel and connected to a battery-operated stimulator system. Direct current with maximal intensity of 1.5 mA with be provided for 20 minutes.
  Arms: Cathodal transcranial direct current stimulation
Device: Sham cathodal transcranial direct current stimulation — Sham stimulation will be performed by the same protocol as active stimulation; however, the device will be switched off 30 seconds after the beginning of stimulation. This way, the patient will experience the same sensations as with active stimulation without receiving actual stimulation.
  Arms: Sham transcranial direct current stimulation

SUMMARY:
Electrophysiological changes that occur in the brains of migraine patients, lead to the activation of nociceptive centers, including a peripheral neural structure, the trigeminal ganglion (TG), which releases pain-inducing peptides and mostly calcitonin gene-related peptide (CGRP). Monoclonal antibodies acting on the CGRP pathway (CGRP-MAbs) are the first drugs specifically designed for migraine, they inhibit CGRP release from the TG without entering the brain. Not all patients experience benefit from CGRP-MAbs treatment. For this reason, associating these drugs with a non-pharmacological treatment that acts centrally, such as transcranial direct current stimulation, could be effective.

The aim of the study is investigating how the migraine preventive treatment with CGRP-MAbs in association with tDCS, is effective to reduce headache days, days of disabling headache, intensity of pain and consumption of acute treatments. Migraine-related disability, quality of life, sleep disturbance and psychological aspects will also be evaluated. Patients will be randomized into two groups, one will receive active tDCS and one sham tDCS. Both patients and investigators will be blind to the treatment administered (double-blind).

Furthermore, will be evalutated the cortical mechanisms involved in migraine by directly modulating brain physiology via repetitive tDCS in patients with migraine on treatment with CGRP-MAbs. To fulfill this aim, we will assess the EEG correlates of the actual effects of the stimulation in a sham-controlled study, providing the EEG indexes linked to the altered and potentially restored cortical dynamics in migraine.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, aged between 40 and 70 years, referring to the Headache Center of the University of L'Aquila;
* a diagnosis of migraine with or without aura according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3; https://ichd-3.org/);
* age at onset of migraine <50 years;
* migraine must have been present for at least ≥ 12 months;
* treated with CGRP-MAbs (erenumab, fremanezumab or galcanezumab) according to clinical practice criteria for 90-180 days since the first subcutaneous administration (this time range was chosen to ensure a stable CGRP pathway inhibition);
* reporting >4 monthly migraine days in the last 30 days of observation despite treatment with CGRP-MAbs;
* able to discriminate between migraine and tension-type headaches;
* written informed consent to participate in the study

Exclusion Criteria:

* any migraine preventive medication other than CGRP-MAbs;
* secondary migraine;
* epilepsy or any other neurologic condition that may be worsened by transcranial electrical stimulation;
* metallic head implants, cardiac pacemaker or any other device that could malfunction or be displaced by electrical stimulation;
* pregnancy or lactation.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Decrease in headache days | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group
Decrease in disabling headache days | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group
Decrease in mean 10-point Visual Analog Scale | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group in the 10-point Visual Analog Scale (0 to 10 points, where 0 means "no pain at all" and 10 "maximum conceivable pain")
Decrease in doses of acute treatment | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group

SECONDARY OUTCOMES:
Decrease in mean modified Migraine Disability Assessment Scale (mMIDAS) score | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group in the modified Migraine Disability Assessment Scale (mMIDAS).
  mMIDAS is a self-administered questionnaire that contains five questions about the headache a patient had in the previous month, assessing the impact of migraine on three domains of daily activity: two questions for paid work or schoolwork, two questions for household work, and one question for family, social and leisure activities. The two questions for each of the first two groups assess, respectively, the number of days off due to headache, and the number of days in which the productivity was reduced by half or more. mMIDAS index is derived from the sum of the answers on the first five questions. This score defines patients in four categories of headache disability: little/none disability if the score is between 0 and 5; mild disability if between 6 and 10; moderate disability if between 11 and 20; and severe disability if greater than 20.
Decrease in mean Headache Impact Test-6 (HIT-6) score | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group
Decrease in mean Short Form Health Survey (SF-36) score | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group
Decrease in mean Pittsburgh Sleep Quality Index (PSQI) score | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group
Decrease in mean Hospital Anxiety and Depression Scale (HADS) score | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group.
  HADS is a scale based upon 14 questions. A score from 0 to 21 is given to both anxiety and depression, where 0-7 scores are normal, 8-10 borderline, and 11-21 abnormal.

OTHER OUTCOMES:
Change in occipital electroencephalographic (EEG) signal power at 8-13 Hz frequency after vs before tDCS | 4 weeks
  Difference between the active tDCS treated group and the sham tDCS treated group

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ornello R, D'Atri A, De Icco R, De Santis F, Rosignoli C, Onofri A, Vaghi G, Cammarota F, Brancaccio C, Corrado M, Bighiani F, Grillo V, Sances G, Corigliano D, Salfi F, Tassorelli C, Ferrara M, Sacco S. Effectiveness of transcranial direct current stimulation and monoclonal antibodies acting on the CGRP as a combined treatment for migraine (TACTIC): Results of a randomized controlled trial. Cephalalgia. 2025 May;45(5):3331024251325567. doi: 10.1177/03331024251325567. Epub 2025 May 19. PMID 40384614
- [Derived] Ornello R, Rosignoli C, Caponnetto V, Pistoia F, Ferrara M, D'Atri A, Sacco S. Effectiveness of Transcranial Direct Current Stimulation and Monoclonal Antibodies Acting on the CGRP as a Combined Treatment for Migraine (TACTIC): Protocol for a Randomized, Double-Blind, Sham-Controlled Trial. Front Neurol. 2022 May 10;13:890364. doi: 10.3389/fneur.2022.890364. eCollection 2022. PMID 35620782